CLINICAL TRIAL: NCT03654417
Title: A Comparison of Pain Perception Using Topical EMLA Cream Versus Lidocaine Injection for Vulvar Biopsy: a Randomized Controlled Trial
Brief Title: Pain Perception During Vulvar Biopsy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: interim analysis produced significant results, so we ended enrollment
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00094298
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Any Condition Requiring Vulvar Biopsy
Keywords: vulvar biopsy
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- EMLA (Active Comparator)
  Interventions: Drug: Lidocaine
- Lidocaine (Active Comparator)
  Interventions: Drug: EMLA

INTERVENTIONS:
Drug: EMLA — Patients undergoing a vulvar biopsy will be randomized to receive EMLA cream or a lidocaine injection as their numbing agent prior to the procedure.
  Arms: Lidocaine
Drug: Lidocaine — Patients undergoing a vulvar biopsy will be randomized to receive EMLA cream or a lidocaine injection as their numbing agent prior to the procedure.
  Arms: EMLA

SUMMARY:
The purpose of this study is to compare pain control during vulvar biopsy following either (1) application of EMLA (a eutectic mixture of local anesthetics lidocaine 2.5% and prilocaine 2.5%) cream or (2) injection of 1% lidocaine. We hypothesize that lidocaine will provide better biopsy analgesia, but the benefit will be offset by the pain of lidocaine injection compared to EMLA application, thus there will not be a significant difference in highest pain scores between the two groups.

DETAILED DESCRIPTION:
Performing minor procedures in-office is essential to gynecologic practices. In-office procedures allow for evaluation and diagnosis of a variety of conditions while avoiding the expense, anesthesia, and time associated with the operating room. Pain and discomfort are frequently associated with these procedures, and ensuring that the patient has the least amount of discomfort is a priority. Very painful or uncomfortable procedures could potentially discourage a patient from returning to clinic or receiving the follow up that they may need. Psychological, physiologic, and social factors influence a patient's experience of pain. Previous studies, though mostly related to first trimester abortion procedures in the office, indicate that the procedure type, anxiety, depression, and general anticipation of pain predict increased pain during in office gynecologic procedures (1-4). A review by Ireland et al., found that a multimodal approach that includes patient counseling with other techniques is most effective in achieving optimum pain control for procedures (5,6).

Vulvar biopsies are associated with significant discomfort, and some form of anesthesia is required. The current standard in our group is to inject local anesthesia prior to vulvar biopsy. However, the injection itself is associated with its own level of pain that is not insignificant, and for many, the anticipation of receiving an injection is anxiety provoking. The use of topical anesthesia in lieu of injection or as pre-injection analgesia is variable.

Several previous studies have examined the use of topical anesthetics in the place of or in addition to injected anesthesia. Drouault et al. compared EMLA cream alone to injected lidocaine alone for pain relief in vulvar biopsy and found that pain associated with administration of anesthesia was significantly less for EMLA cream, but better biopsy analgesia was obtained with injected anesthesia. The study considered combined pain scores for both groups for the overall procedure (anesthesia + biopsy), it comments that the combined scores were lower for the EMLA group but failed to reach statistical significance. The study ultimately concluded that EMLA is the less painful procedure to obtain anesthesia and that it can be used as an alternative to injection for biopsies of the genital mucosa (7). This prior study did not compare the highest pain score between groups. Consideration of the highest pain score allows us to assess whether the injection of lidocaine could result in causing more pain than the biopsy itself using EMLA cream alone for anesthesia. Further, the study did not assess the subjects' or the providers' perception of the tolerability and acceptability of performing the procedure using either method. This is an important factor in any in office procedure

EMLA cream is the most extensively studied topical anesthetic. It is FDA approved for use as a topical anesthetic on the genital mucous membranes for superficial, minor surgery. EMLA cream requires between 7-10 minutes of absorption time on the genital mucosa for analgesic effect, with variable duration of analgesia following, usually around 15-20 minutes (9). There is a highly variable absorption rate for EMLA cream depending on the characteristics of the epithelium upon which it is applied as well as the duration and surface area of cream applied. On hair-bearing non-mucosal surfaces it can require 60 minutes of application time to obtain analgesic affect (10). The vulvar area is unique in that it contains both mucosal and non-mucosal and hair-bearing surfaces; this could greatly affect the absorption of EMLA and therefore affect analgesia. For this reason, we will exclude from the study patients requiring vulvar biopsy on hair bearing portion of the vulva.

Several previous studies have examined the use of topical anesthetics in the place of or in addition to injected anesthesia. Drouault et al. compared EMLA cream to injected lidocaine as described above. The study found that pain associated with administration of anesthesia was significantly less for EMLA cream, but better biopsy analgesia was obtained with injected anesthesia. However, there were some limitations to this study also noted above, that we plan to expand and improve upon with the current study.

Zilbert and Lewandoswki studied pre-treatment with EMLA cream prior to anesthesia injection and found that pain was decreased by 50% in patients pretreated compared to placebo prior to lidocaine injection.

Van den Berg studied application of EMLA alone versus lidocaine injection alone in punch biopsies and electrocoagulation of genital warts in men. The study found that in the punch biopsy cohort that the total pain scores (application of EMLA + biopsy versus injection of lidocaine + biopsy) were less for the EMLA group than the injected lidocaine group and the difference was statistically significant (11).

With its FDA approval for use as a topical anesthetic on the genital mucous membranes for superficial, minor surgery, it can be considered a standard of care to use EMLA for anesthesia prior to biopsy as an alternative to injection of lidocaine (10)

As there are no studies that consider the subjects' or the providers' perception of the acceptability or the tolerability of the procedure, this will be novel data for vulvar biopsy. However, acceptability and tolerability have been assessed in other procedural settings, such as in office endoscopic procedures, in which BS-11, a validated 11 point scale, is used to assess pain, anxiety, acceptability, tolerability, and levels of other procedure related symptoms (12-13).

ELIGIBILITY:
Inclusion Criteria:

* Females above age 18 presenting to Duke Gynecology Oncology clinic for vulvar biopsy
* Able to provide informed consent in English and agree to the risks of the study

Exclusion Criteria:

* Not able to provide informed consent
* Vulvar biopsy on a hair bearing surface

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Havrilesky, MD, Principal Investigator — Duke University
Locations (1):
- Duke Univeristy, Durham, North Carolina, United States

REFERENCES:
- [Derived] Williams LK, Weber JM, Pieper C, Lorenzo A, Moss H, Havrilesky LJ. Lidocaine-Prilocaine Cream Compared With Injected Lidocaine for Vulvar Biopsy: A Randomized Controlled Trial. Obstet Gynecol. 2020 Feb;135(2):311-318. doi: 10.1097/AOG.0000000000003660. PMID 31923074

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EMLA | Lidocaine
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EMLA | Lidocaine | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [46 to 74] | 58.5 [51 to 65] | 60 [51 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 18 | 18 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 12 | 9 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Highest Pain Score
Description: The highest pain score recorded (at time of numbing or at time of biopsy) controlled for baseline pain
  title: Please slide the tab along the line below to indicate pain in the area of your vulva (external genitalia) during numbing OR biopsy min: 0 (no pain) max: 100 (worst pain imaginable)
Time Frame: no more than 5 minutes after numbing or 5 minutes after biopsy
Measure: Median (Inter-Quartile Range); unit: units on a scale (mm)
Arm/Group | EMLA | Lidocaine
Number analyzed (Participants) | 19 | 18
units on a scale (mm) | 20 [5 to 50] | 56.5 [26 to 80]

2. Secondary Outcome: Pain During Biopsy as Measured by a Pain Scale
Description: self-reported level of pain following the biopsy
  title: Please slide the tab along the line below to indicate pain in the area of your vulva (external genitalia) during biopsy min: 0 (no pain) max: 100 (worst pain imaginable)
Time Frame: No more than 5 minutes after receiving the biopsy
Measure: Median (Inter-Quartile Range); unit: units on a scale (mm)
Arm/Group | EMLA | Lidocaine
Number analyzed (Participants) | 19 | 18
units on a scale (mm) | 6 [1 to 50] | 3 [0 to 15]

3. Secondary Outcome: Baseline Vulvar Pain
Description: self-reported level of vulvar pain immediately prior to the start of the procedure title: Please slide the tab along the line below to indicate pain in the area of your vulva (external genitalia) during biopsy min: 0 (no pain) max: 100 (worst pain imaginable)
Time Frame: no more than 30 minutes prior to procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale (mm)
Arm/Group | EMLA | Lidocaine
Number analyzed (Participants) | 19 | 18
units on a scale (mm) | 0.0 [0.0 to 5.0] | 0.0 [0.0 to 3.0]

4. Secondary Outcome: Anxiety Before the Procedure as Measured by an Anxiety Scale
Description: self-reported level of anxiety immediately prior to the start of the procedure
  title: Slide the tab along the line below to indicate how nervous you feel about the procedure you are about to have min: 0 (not nervous) max: 100 (very nervous)
Time Frame: No more than 30 minutes before the procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale (mm)
Arm/Group | EMLA | Lidocaine
Number analyzed (Participants) | 19 | 18
units on a scale (mm) | 19 [0.0 to 31.0] | 31.5 [12.0 to 61.0]

5. Secondary Outcome: Generalized Anxiety Disorder 7-item (GAD-7) Score for Baseline Anxiety
Description: Self-reported anxiety score meant to assess a patient's baseline level of anxiety. The score ranges from 0 (minimal anxiety) to 21 (severe anxiety).
Time Frame: no more than 30 minutes before the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | EMLA | Lidocaine
Number analyzed (Participants) | 19 | 18
Participants
  Minimal Anxiety (0-4) | 13 | 11
  Mild Anxiety (5-9) | 5 | 5
  Moderate Anxiety (10-14) | 0 | 1
  Severe Anxiety (15-21) | 1 | 1

6. Secondary Outcome: Acceptance of the Procedure as Measured by a Satisfaction Scale
Description: self-reported acceptance of the procedure meant to assess a patient's acceptability through a scale
  title: Please slide the tab along the line below to indicate, overall, how acceptable the procedure performed today was min: 0 (completely acceptable) max: 100 (not at all acceptable)
Time Frame: up to 30 minutes after the procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale (mm)
Arm/Group | EMLA | Lidocaine
Number analyzed (Participants) | 19 | 18
units on a scale (mm) | 0 [0 to 18] | 10.5 [1 to 33]

7. Secondary Outcome: Tolerance of Procedure as Measured by a Satisfaction Scale
Description: self-reported tolerance of the procedure meant to assess a patient's tolerance through a scale
  Title: Please slide the tab along the line below to indicate, overall, how you would rate the experience of your biopsy procedure today Min: 0 (I could easily handle having this procedure again) Max: 100 (I could never have this procedure done again)
Time Frame: Up to 30 minutes after the procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale (mm)
Arm/Group | EMLA | Lidocaine
Number analyzed (Participants) | 19 | 18
units on a scale (mm) | 2 [0 to 17] | 17 [5 to 38]

8. Secondary Outcome: Provider's Opinion of Subject Tolerance as Measured by a Scale
Description: provider-reported measure of how well they believe the patient tolerated the procedure
  title: Overall, how well did the subject tolerate the procedure today? min: 0 (well tolerated) max: 100 (poorly tolerated)
Time Frame: Up to 30 minutes after the procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale (mm)
Arm/Group | EMLA | Lidocaine
Number analyzed (Participants) | 19 | 18
units on a scale (mm) | 3 [0 to 19] | 15 [9 to 27]

9. Secondary Outcome: Provider's Overall Satisfaction With the Procedure as Measured by a Scale
Description: provider-reported measure of how well they believe the procedure went
  title: Overall, how satisfied are you with the procedure performed today? min: 0 (completely satisfied) max: 100 (not at all satisfied)
Time Frame: Up to 30 minutes after the procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale (mm)
Arm/Group | EMLA | Lidocaine
Number analyzed (Participants) | 19 | 18
units on a scale (mm) | 3 [0 to 18] | 9.5 [3 to 18]

10. Post Hoc Outcome: Possible Pathologic Changes Associated With EMLA Cream Application
Description: To address the concern that EMLA might induce pathologic changes that could result in altered diagnosis, pathologist independent from initial diagnostic read will re-evaluate tissue slides and look for the previously described EMLA induced pathologic changes (pallor, necrosis, spongiosis, basophilic granules, acantholysis, clefting, papillary dermal edema). Pathologist will be blinded to whether or not patient received EMLA cream for biopsy. They will provide a score for all specimens that will be used to analyse any pathologic differences between patients exposed to EMLA and those not exposed to EMLA.
Time Frame: retrospective
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 30 minutes after the procedure
Arm/Group | EMLA | Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

LIMITATIONS AND CAVEATS:
unblinded patients and providers, prior experience with vulvar biopsy may be biasing, pre-procedure anxiety may be biased because posed after randomization, no gold standard for pain assessment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Informed Consent Form (2018-11-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT03654417/ICF_000.pdf
  • Study Protocol (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT03654417/Prot_001.pdf
  • Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT03654417/SAP_002.pdf